CLINICAL TRIAL: NCT02343354
Title: The MoMMii Study: Effects of a Multimodal Diabetes Prevention Intervention on Families With a History of Gestational Diabetes
Brief Title: The MoMMii Study. Diabetes Prevention Intervention on Families With Past Gestational Diabetes
Acronym: MoMMii
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: The Lawson Foundation (Other)
Responsible Party: Principal Investigator, Kaberi Dasgupta, MD, MSc, FRCP (C), Physician-Scientist and Director of Clinical Epidemiology, MUHC, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GRT 2014-35
Record Dates: First submitted 2015-01-15; First posted 2015-01-22 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Gestational Diabetes Mellitus With Baby Delivered
Keywords: behavioural; diabetes prevention; physical activity; healthy eating; gestational diabetes
MeSH Terms: conditions — Motor Activity; Diabetes, Gestational | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutrition/physical activity intervention (Experimental): There will be five in-person group sessions (3 to 4 weeks appart) with on-site child care. Sessions will include preparation of a healthy meal (hands-on) and discussions of mindful eating, balanced meals, portion sizes, and preparing food at home, under a dietitian's supervision. Sessions will also include a one-hour physical activity information/practice session with a kinesiologist. Participants will track daily step counts with a pedometer and aim to eventually reach more than 10,000 steps/day. They will also receive instruction and demonstration from a kinesiologist of some simple resistance exercises they may perform at home. Between sessions, participants will receive advice and support through a study-specific website, telephone calls and phone applications.
  Interventions: Behavioral: Nutrition/physical activity intervention

INTERVENTIONS:
Behavioral: Nutrition/physical activity intervention — Please see arm description
  Other Names: Lifestyle intervention; Diabetes prevention intervention

SUMMARY:
Women with gestational diabetes (GDM) have increased risk of developing type 2 diabetes; their children show more insulin resistance and diabetes compared to offspring of mother without diabetes in pregnancy. An increased diabetes risk is also observed among partner of adult with prediabetes/type 2 diabetes. The investigators have pilot-tested a program for diabetes risk reduction among women within 5 years of a GDM pregnancy (MoMM program). The investigators are now enhancing the program to engage directly the partner (MoMMii program).

In MoMMii, 66 couples with a history GDM in the mother will participate in a multimodal diabetes prevention program that includes healthy meal preparation training, discussion of eating and physical activity behaviours and developing home environments that facilitate healthy habits, pedometer-based step count monitoring, and participation in family-based activities (frisbee, soccer) as well as individual exercise (e.g., use of exercise equipment, floor resistance exercises). Participants will be encouraged to communicate between sessions with study personnel and with one another to create a between family support network. All mothers and fathers will participate in five sessions over six months. The investigators will examine changes in health-related behaviours, blood pressure, glucose levels, and insulin sensitivity/resistance in both mothers and fathers.

DETAILED DESCRIPTION:
The primary goal of the project is to determine if, among families with a history of gestational diabetes mellitus (GDM) in the mother in the prior five years, a family-based multimodal health behaviour intervention (group cooking and eating/physical activity counselling, telephone-based app and text support, building of peer and within-family social support for health behaviour change) will lead to reductions in post 75g glucose load serum glucose values in mothers and fathers. The previous MoMM pilot study demonstrated an 8% reduction in mothers, similar in magnitude to that observed in a large diabetes prevention trial conducted among adults with impaired glucose tolerance (Tuomieltho et al, N Engl J Med 2001). MoMMii will ascertain if expansion to a family-based approach amplifies effects in mothers and demonstrates impact in fathers and children. Thus, MoMMii will shift the focus from the mother to the family. A systematic review and meta-analysis showed diabetes risk to be shared between spouses (Leong et al, BMC Medicine, 2014). GDM also confers higher risk for insulin resistance and overweight in offspring. Thus, this project plans to create a collaborative home environment that facilitates choices consistent with diabetes prevention for all family members. Sixty-six families will be recruited through GDM clinics at McGill University Health Centre and other centres. Five in-person sessions (meal preparation training, eating and physical activity counselling) will take place once a month at the PERFORM Centre, Concordia University. Each session will involve discussion of strategies to achieve healthy eating, hands-on meal preparation, and group-based physical activity. Sessions will engage couples as well as mothers and fathers separately. 'Healthy living' concepts will be integrated into the on-site childcare structure (meal preparation, games, videos). The intervention team will include a dietitian and kinesiologist. A health coach will facilitate networking among participating families and development of lay group leaders to sustain health behaviour changes between sessions and post program. Outcomes will be evaluated in mothers, fathers (e.g., fasting and post load glucose and insulin resistance measures, fruit/vegetable intake, step counts, eating behaviours, blood pressure) and offspring (dietary/physical activity habits).

ELIGIBILITY:
Inclusion Criteria:

1. Prior history of gestational diabetes in the mother
2. Ability to speak and read English or French

Exclusion Criteria:

1. Other forms of diabetes (e.g., type 1 diabetes, type 2 diabetes)
2. Current use of antihyperglycemic medication
3. Pregnancy or attempting to become pregnant
4. Chronic condition/ medications that could impact weight (e.g. malignancy, weight loss medications, anti-depressants)
5. Current smoker

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2014-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in post 75 gram glucose load 2-hour glucose value in mothers and fathers | 20-24 weeks
  Following an overnight fast and venous blood sampling for fasting glucose, a 75 gram glucose solution will be consumed by the participant and two hours later, venous blood will be sampled for a repeat serum glucose assay. The pre-intervention value will be subtracted from the post-intervention value to compute the change during the intervention.

SECONDARY OUTCOMES:
Change in fruit and vegetable consumption in mothers and fathers | 20-24 weeks
  Estimates of consumption based on food frequency questionnaire data completed by mothers and fathers. The pre-intervention value will be subtracted from the post-intervention value to compute the change during the intervention.
Change in physical activity in mothers and fathers | 20-24 weeks
  Daily physical activity assessed by accelerometers and pedometer-based step counts in mothers and fathers. The pre-intervention value will be subtracted from the post-intervention value to compute the change during the intervention.
Change in insulin resistance measure (HOMA-IR) in mothers and fathers | 20-24 weeks
  Homeostatic Assessment of insulin resistance (HOMA-IR) calculated with fasting glucose and fasting insulin values. The pre-intervention value will be subtracted from the post-intervention value to compute the change during the intervention.
Change in insulin sensitivity measure (ISI 0,120) in mothers and fathers | 20-24 weeks
  Using the ratio of the serum insulin levels at the 0 minute and 120-minute time points, the insulin sensitivity index (ISI 0, 120), another marker of insulin resistance, will be calculated as proposed in Gutt M, Davis CL, Spitzer SB, Llabre MM, Kumar M, Czarnecki EM et al. Validation of the insulin sensitivity index (ISI(0,120)): comparison with other measures. Diabetes Res Clin Pract 2000; 47(3):177-184. The pre-intervention value will be subtracted from the post-intervention value to compute the change during the intervention.
Change in fasting glucose in mothers and fathers | 20-24 weeks
  Following an overnight fast, venous blood will be sampled for assessment of fasting glucose. The pre-intervention value will be subtracted from the post-intervention value to compute the change during the intervention.
Change in fasting insulin in mothers and fathers | 20-24 weeks
  Following an overnight fast, venous blood will be sampled for assessment of fasting insulin. The pre-intervention value will be subtracted from the post-intervention value to compute the change during the intervention.
Change in systolic blood pressure in mothers and fathers | 20-24 weeks
  Systolic blood pressure will assessed with the participant seated in a quiet room with the arm supported. Measurements will be taken with an automated device at 1-minute intervals for 6 sequential measurements. The latter 5 measurements will be averaged. The pre-intervention (average) systolic blood pressure will be subtracted from the post-intervention (average) systolic blood pressure for computation of the change in systolic blood pressure.
Change in diastolic blood pressure in mothers and fathers | 20-24 weeks
  Diastolic blood pressure will assessed with the participant seated in a quiet room with the arm supported. Measurements will be taken with an automated device at 1-minute intervals for 6 sequential measurements. The latter 5 measurements will be averaged. The pre-intervention (average) diastolic blood pressure will be subtracted from the post-intervention (average) diastolic blood pressure for computation of the change in systolic blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Kaberi Dasgupta, MD, MSc, Principal Investigator — McGill University and McGill University Health Centre
Locations (1):
- McGill University Health Centre - Royal Victoria Hosptial, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brazeau AS, Meltzer SJ, Pace R, Garfield N, Godbout A, Meissner L, Rahme E, Da Costa D, Dasgupta K. Health behaviour changes in partners of women with recent gestational diabetes: a phase IIa trial. BMC Public Health. 2018 May 2;18(1):575. doi: 10.1186/s12889-018-5490-x. PMID 29716559
- [Background] Brazeau AS, Leong A, Meltzer SJ, Cruz R, DaCosta D, Hendrickson-Nelson M, Joseph L, Dasgupta K; MoMM study group. Group-based activities with on-site childcare and online support improve glucose tolerance in women within 5 years of gestational diabetes pregnancy. Cardiovasc Diabetol. 2014 Jun 30;13:104. doi: 10.1186/1475-2840-13-104. PMID 24981579
- [Background] Leong A, Rahme E, Dasgupta K. Spousal diabetes as a diabetes risk factor: a systematic review and meta-analysis. BMC Med. 2014 Jan 24;12:12. doi: 10.1186/1741-7015-12-12. PMID 24460622
- [Background] Dasgupta K, Da Costa D, Pillay S, De Civita M, Gougeon R, Leong A, Bacon S, Stotland S, Chetty VT, Garfield N, Majdan A, Meltzer S. Strategies to optimize participation in diabetes prevention programs following gestational diabetes: a focus group study. PLoS One. 2013 Jul 4;8(7):e67878. doi: 10.1371/journal.pone.0067878. Print 2013. PMID 23861824
- See also: MoMM pilot study — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4227099/